CLINICAL TRIAL: NCT01743781
Title: The Impact of Multimedia Education on Uptake of Comprehensive Eye Examination in Rural Southern China:A Randomized, Controlled Trial
Brief Title: Uptake of Comprehensive Eye Examination Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Orbis (Other); The World Diabetes Foundation (Other)
Responsible Party: Principal Investigator, Congdon Nathan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZOC-CREST2
Record Dates: First submitted 2012-11-21; First posted 2012-12-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Glaucoma; Diabetic Retinopathy
Keywords: comprehensive eye examination; acceptance; glaucoma; diabetic retinopathy
MeSH Terms: conditions — Glaucoma; Diabetic Retinopathy | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental): view a 10-minute informational video about comprehensive eye examination
  Interventions: Behavioral: video
- control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: video — view a 10-minute informational video about comprehensive eye examination
  Arms: intervention group

SUMMARY:
1. To evaluate a educational intervention promoting acceptance of comprehensive eye examination in rural Guangdong.
2. To evaluate the impact of acceptance of comprehensive eye examination in rural Guangdong.

DETAILED DESCRIPTION:
A comprehensive eye examination includes visual acuity, slitlamp exam, pupil exam, intraocular pressure, gonioscope lens and 90D lens with slitlamp exam fundus. A number of eye diseases are irreversible at on early stage. Both glaucoma and diabetic retinopathy(DR)are frequently asymptomatic until significant, often-irreversible, damage to the vision has already occurred. It has been estimated that only 10% of persons in India with glaucoma are diagnosed, and the Handan Eye Survey reports that only 10% of persons with diabetes in rural areas of China have received diabetic eye care. In order to deliver effective care for DR and glaucoma in areas with limited resources, education of patients and interventions to promote compliance among patients will both be needed.

ELIGIBILITY:
Inclusion Criteria:

* age ≥40 years who have never had a comprehensive eye examination

Exclusion Criteria:

* inability to join informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The acceptance rate of comprehensive eye examination in both groups | 1 day
  acceptance rate of comprehensive eye examination

SECONDARY OUTCOMES:
knowledges of eye disease and attitude of eye examination | 1 day
  knowledges of eye disease and attitude of eye examination

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD,MPH, Principal Investigator — Sun yat-sen university, Zhongshan Ophthalmic Center; Mingguang He, MD,PHD, Principal Investigator — Sun Yat-sen University,Zhongshan Ophthalmic Center; Aihua Dan, MD, Principal Investigator — Sun Yat-sen University,Zhongshan Ophthalmic Center
Locations (1):
- 54 Xianlie Rd, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Dan A, Raubvogel G, Chen T, Ye T, Jin L, Xiao B, Sanchez A, Congdon N. The Impact of Multimedia Education on Uptake of Comprehensive Eye Examinations in Rural China: A Randomized, Controlled Trial. Ophthalmic Epidemiol. 2015;22(4):283-90. doi: 10.3109/09286586.2015.1056812. PMID 26218111